CLINICAL TRIAL: NCT04078737
Title: Clopidogrel With Aspirin in High-risk Patients With Acute Non-disabling Cerebrovascular Events II
Acronym: CHANCE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017ZX09304018001; NCT04952311 (obsolete NCT alias)
Record Dates: First submitted 2019-07-08; First posted 2019-09-06 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Stroke; Transient Ischemic Attack
Keywords: stroke; transient ischemic attack; acute treatment; acute non-disabling cerebrovascular event; clopidogrel; ticagrelor; clopidogrel combined with ASA; ticagrelor combined with ASA; recurrence of stroke and other vascular events; CYP2C19 loss-of-function allele(s) carrier
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor plus Aspirin Group (Experimental): Ticagrelor of loading dosing of 180mg followed by 90mg bid for 3 months plus aspirin of loading dose of 75-300mg followed by 75mg daily for 21 days
  Interventions: Drug: Ticagrelor and Aspirin
- Clopidogrel plus Aspirin Group (Active Comparator): Clopidogrel of loading dosing of 300mg followed by 75mg daily for 3 months plus aspirin loading dose of 75-300mg followed by 75mg daily for 21 days
  Interventions: Drug: Clopidogrel and Aspirin

INTERVENTIONS:
Drug: Ticagrelor and Aspirin — Day of randomization:
  Day1:Ticagrelor 180mg; placebo of clopidogrel 300mg; aspirin 75-300mg (open label) Day2-21st: Ticagrelor 90mg bid/day; placebo of clopidogrel 75mg; aspirin 75mg (open label) Day 22nd-3 months:Ticagrelor 90mg bid/day; placebo of clopidogrel 75mg
  Arms: Ticagrelor plus Aspirin Group
Drug: Clopidogrel and Aspirin — Day of randomization:
  Day 1: Clopidogrel 300mg; placebo of ticagrelor 180mg; aspirin 75-300mg (open label) Day2-21st: Clopidogrel 75mg/day; placebo of ticagrelor 90mg bid/day; aspirin 75mg (open label) Day 22nd-3 months:Clopidogrel 75mg; placebo of ticagrelor 90mg bid/day
  Arms: Clopidogrel plus Aspirin Group

SUMMARY:
The primary objective of this trial is to assess the effects of ticagrelor plus aspirin versus clopidogrel plus aspirin on reducing the 3-month risk of any stroke (both ischemic and hemorrhagic, primary outcome) when initiated within 24 hours of symptom onset in CYP2Y19 LOF alleles carriers with TIA or minor stroke.

DETAILED DESCRIPTION:
According to the Global Burden of Disease(GBD) Study 2016, China bears the greatest lifetime risk of stroke from 25-year-age onward. Minor ischemic events, including minor stroke and TIA, were major parts of stroke manifestations. Events (CHANCE) has shown that 21-day dual antiplatelet therapy (clopidogrel and aspirin) compared to aspirin alone which initiated within 24 hours after symptoms onset would reduce 32% risk of stroke recurrence within 90 day, but not in carriers of CYP2C19 loss-of-function (LOF) alleles. The primary purpose of this study is to compare ticagrelor plus aspirin with clopidogrel plus aspirin on reducing the 3-month risk of any stroke (both ischemic and hemorrhagic, primary outcome) when initiated within 24 hours of symptom onset in CYP2Y19 LOF alleles carriers with TIA or minor stroke.

Both intent analysis (ITT) and compliance program set (PPS) were used for analysis.

We will use Kaplan-Meier estimates of the cumulative risk of stroke (ischemic or hemorrhagic) event during maximum 90-day follow-up, with hazards ratios and 95% CI calculated using Cox proportional hazards methods and the log-rank test to evaluate the treatment effect. All statistics will be 2-sided with P<0.05 considered significant, accounting for interim analyses.

All patients who received study drugs and with at least one safety follow-up record will be included in the safety population. The data for safety evaluation included adverse reactions observed during the trial and changes in laboratory data before and after treatment.

ELIGIBILITY:
Inclusion Criteria

1. 40 years or older than 40 years；
2. Acute cerebral ischemic event due to：

   * Acute non-disabling ischemic stroke (NIHSS≤3 at the time of randomization)or，
   * TIA with moderate-to-high risk of stroke (ABCD2 score ≥ 4 at the time of randomization)；
3. Can be treated with study drug within 24 hours of symptoms onset*(*Symptom onset is defined by the "last seen normal" principle)；
4. CYP2C19 loss-of-function allele carriers；
5. Informed consent signed.

Exclusion Criteria

1. Malformation, tumor, abscess or other major non-ischemic brain disease (e.g., multiple sclerosis) on baseline head CT or MRI.
2. Isolated or pure sensory symptoms (e.g., numbness), isolated visual changes, or isolated dizziness/vertigo without evidence of acute infarction on baseline head CT or MRI.
3. Iatrogenic causes (angioplasty or surgery) of minor stroke or TIA.
4. Preceding moderate or severe dependency (modified Rankin scale [mRS] score 3-5).
5. Contraindication to clopidogrel, ticagrelor or aspirin

   * Known allergy
   * Severe renal (creatinine exceeding 1.5 times of the upper limit of normal range) or hepatic (ALT or AST > twice the upper limit of normal range) insufficiency
   * Severe cardiac failure (NYHA level: III to IV)
   * History of hemostatic disorder or systemic bleeding
   * History of thrombocytopenia or neutropenia
   * History of drug-induced hematologic disorder or hepatic dysfunction
   * Low white blood cell (<2×109/L) or platelet count (<100×109/L)
6. Hematocrit (HCT) <30%
7. Clear indication for anticoagulation (presumed cardiac source of embolus, e.g., atrial fibrillation, prosthetic cardiac valves known or suspected endocarditis)
8. History of intracranial hemorrhage or amyloid angiopathy
9. History of aneurysm (including intracranial aneurysm and peripheral aneurysm)
10. History of asthma or COPD (chronic obstructive pulmonary disease)
11. High-risk for bradyarrhythmia (first-degree or second-degree AV block caused by sinus node disease, and brady-arrhythmic syncope without pacemaker)
12. History of hyperuricemia nephropathy
13. Anticipated requirement for long-term (>7 days) non-steroidal anti-inflammatory drugs (NSAIDs)
14. Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
15. Scheduled for surgery or interventional treatment requiring study drug cessation
16. Severe non-cardiovascular comorbidity with life expectancy < 3 months
17. Inability to understand and/or follow research procedures due to mental, cognitive, or emotional disorders
18. Dual antiplatelet treatment (or more than two antiplatelet agents) in 72 hours before randomization
19. Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anti coagulation
20. Intravenous thrombolytic therapy (such as intravenous rtPA) or mechanical thrombectomy within 24 hours prior to randomization
21. Gastrointestinal bleed within 3 months or major surgery within 30 days
22. Diagnosis or suspicious diagnosis of acute coronary syndrome
23. Participation in another clinical study with an experimental product during the last 30 days
24. Currently receiving an experimental drug or device
25. Pregnant, currently trying to become pregnant, or of child-bearing potential and not using birth control

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6412 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Any new stroke events (ischemic stroke or hemorrhagic stroke) within 3 months | 3 months after randomization
  The aim is to assess the effects of ticagrelor plus aspirin versus clopidogrel plus aspirin on reducing the 3-month risk of any stroke (both ischemic and hemorrhagic, primary outcome) when initiated within 24 hours of symptom onset in CYP2Y19 LOF alleles carriers with TIA or minor stroke.

SECONDARY OUTCOMES:
Any new stroke events within 30 days and 1 year | 30 days and 1 year after randomization
  Percentage of patients with the 30 days and 1 year new stroke events (ischemic stroke/ hemorrhagic stroke) as a cluster and evaluated individually.
New clinical vascular events including stroke, TIA, myocardial infarction, and vascular deaths within 3 months and 1 year | 3 months and 1 year after randomization
  Percentage of patients with the 3 months and 1 year new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ TIA/ myocardial infarction/vascular death)
New ischemic stroke within 3 months and 1 year | 3 months and 1 year after randomization
  Percentage of patients with the 3 months and 1 year new ischemic stroke will be evaluated.
Disabling stroke (Modified Rankin Scale score, mRS>1) at 3 months and 1 year | 3 months and 1 year after randomization
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome. (dead).
Incidence and severity of recurrent stroke and TIA during follow-up to 3 months and 1-year | 3 months and 1 year after randomization
  (Severity is measured using a six-level ordered categorical scale that incorporates the mRS: fatal stroke/severe non-fatal stroke [mRS 4 or 5]/moderate stroke [mRS 2 or 3]/mild stroke [mRS 0 or 1]/TIA/no stroke-TIA).
Neurological impairment at 3 months (NIHSS increased≥4 from baseline) | 3 months after randomization
  The National Institutes of Health Stroke Scale (NIHSS) score classifies neurologic deficit from 0 (no deficit) to 42 (most severe).
Quality of Life (EuroQol EQ-5D scale) at 3 months and at 1 year | 3 months and 1 year after randomization
  Further efficacy exploratory analysis:Quality of Life (EuroQol EQ-5D scale). We will use the EQ-5D-5L scale to evaluate the quality of life. EQ-5D-5L is a standardized instrument for measuring generic health status. It has been widely used in population health surveys, clinical studies, economic evaluation and in routine outcome measurement in the delivery of operational healthcare. The EQ-5D-5L has five domain scales (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and five levels for each domain.
Stratified analysis | 3 months and 1 year after randomization
  The influence on treatment effect of age, gender, Body Mass Index (BMI), index event type (TIA vs. minor stroke), time from index event to randomization, etiology subtype, diabetes mellitus, hypertension, type of LOF allele, previous ischemic stroke or TIA, prior antiplatelet therapy, prior statin therapy, prior smoking status, and symptomatic intracranial and extracranial artery stenosis will be evaluated in subgroup analyses.

OTHER OUTCOMES:
Moderate and severe bleeding events according to the GUSTO criteria | 3 months after randomization
  Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage.
Moderate and severe bleeding events according to the GUSTO criteria | 1 year after randomization
  Severe bleeding incidence (GUSTO definition), including fatal bleeding and symptomatic intracranial hemorrhage.
All bleeding events | 3 months and 1 year after randomization
  All bleeding events (severe/moderate bleeding and intracranial hemorrhage)
Total mortality | 3 months and 1 year after randomization
  Total mortality
Incidence symptomatic intracranial hemorrhagic events | 3 months and 1 year after randomization
  Incidence symptomatic intracranial hemorrhagic events
Adverse events | 3 months and 1 year after randomization
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, M.D, Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (214):
- China (214):
  - Anqing Municipal Hospital, Anqing, Anhui
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Chaoyang Hospital, Capital MedicalUniversity（west Hospital）, Beijing, Beijing Municipality
  - Beijing Tian tan Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi Airport Hospital, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Beijing, Beijing Municipality
  - Beijing Coal Group Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing People's Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Sanbo Chang 'an Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing Fifth People's Hospital, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - People's Hospital of Rongchang District, Chongqing,, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Chongqing Kaizhou District People's Hospital, Chongqing, Chongqing Municipality
  - Chongqing Fuling Central Hospital, Chongqing, Chongqing Municipality
  - Chongqing Nanchuan District People's Hospital, Chongqing, Chongqing Municipality
  - Xiushan Tujia and Miao Autonomous County People's Hospital, Chongqing, Chongqing Municipality
  - The Third Affiliated Hospital of Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian
  - Fuzhou Second Hospital, Fuzhou, Fujian
  - Sanming First Hospital Affiliated to Fujian Medical University, Sanming, Fujian
  - Wuwei People's Hospital, Wuwei, Gansu
  - Zhangye People's Hospital Affiliated to Hexi College, Zhangye, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital Of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The first Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Guiyang Second People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan West Central Hospital, Danzhou, Hainan
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei Medical University, Baoding, Hebei
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - Hejian People's Hospital, Hejian, Hebei
  - HaLixun InternationalPeace Hospital, Hengshui, Hebei
  - Hengshui fourth People Hospital（Department of Neurology ward 2）, Hengshui, Hebei
  - The Fourth People's Hospital of Hengshui City（Department of Neurology ward 1）, Hengshui, Hebei
  - The Second Hospitalof Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Second Central Hospital of Baoding, Zhuozhou, Hebei
  - Daqing Oilfield Gengeal Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Harbin Medical University（Department of Neurology ward 1）, Harbin, Heilongjiang
  - The Second Hospital of Harbin Medical University（Department of Neurology ward ）, Harbin, Heilongjiang
  - The First Affiliated Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Hongqi Hospital affiliated to Mudanjiang Medical University, Mudanjiang, Heilongjiang
  - Qiqihar Rongjian Institute of Stroke Prevention and Treatment, Qiqihar, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Changge People's Hospital, Jianshe, Henan
  - Xiuwu County People's Hospital, Jiaozuo, Henan
  - Jiyuan People's Hospital, Jiyuan, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - weishi county Central Hospital, Kaifeng, Henan
  - Luohe Central Hospital, Luohe, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - The first Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Luoyang New District People's Hospital, Luoyang, Henan
  - Pingdingshan First People's Hospital, Pingdingshan, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Shangqiu Fourth People's Hospital, Shangqiu, Henan
  - Suixian county Hospital of Traditional Chinese Medicine, Shangqiu, Henan
  - Xingyang People's Hospital, Xingyang, Henan
  - The first Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan
  - Gongyi People's Hospital, Zhengzhou, Henan
  - Zhoukou Yongshan Hospital, Zhoukou, Henan
  - Zhumadian Hospital of Traditional Chinese Medicine, Zhumadian, Henan
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - First hospital of Changsha city, Changsha, Hunan
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - Fourth People's Hospital of Chenzhou, Chenzhou, Hunan
  - The First Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Loudi City Central Hospital, Loudi, Hunan
  - shaoyang Central Hospital, Shaoyang, Hunan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Yueyang Second People's Hospital, Yueyang, Hunan
  - The first Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Baotou CentralHospital, Baotou, Inner Mongolia
  - The second Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Wuyuan County People's Hospital, Bayan Nur, Inner Mongolia
  - Hulun Buir People's Hospital, Buri, Inner Mongolia
  - Chifeng City Hospital, Chifeng, Inner Mongolia
  - Affiliated Hospital of Chifeng University, Chifeng, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia
  - Huaian Hospital of Traditional Chinese Medicine, Huai'an, Jiangsu
  - Lianshui County People's Hospital, Huai'an, Jiangsu
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Gulou Hospital, Nanjing, Jiangsu
  - BenQ Hospital affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Fourth Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Jiangbei People's Hospital, Nanjing, Jiangsu
  - Nanjing Gaochun People's Hospital, Nanjing, Jiangsu
  - Nantong 6th People's Hospital, Nantong, Jiangsu
  - Nantong Hospital of Traditional Chinese Medicine, Nantong, Jiangsu
  - The Third People's Hospital in Tongzhou District, Nantong, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Nantong First People's Hospital, Nantong, Jiangsu
  - Nantong Second People's Hospital, Nantong, Jiangsu
  - Nantong Fourth People's Hospital, Nantong, Jiangsu
  - Nantong Third People's Hospital, Nantong, Jiangsu
  - Tongzhou District People's Hospital of Nantong City, Nantong, Jiangsu
  - Rudong County People's Hospital, Nantong, Jiangsu
  - Rugao People's Hospital, Nantong, Jiangsu
  - Hai 'an People's Hospital, Nantong, Jiangsu
  - Tongzhou District 8th People's Hospital of Nantong City, Nantong, Jiangsu
  - Siyang County People's Hospital, Suqian, Jiangsu
  - Siyang Kangda Hospital, Suqian, Jiangsu
  - Suqian People's Hospital, Suqian, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Xinghua People's Hospital, Taizhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Yixing People's Hospital, Wuxi, Jiangsu
  - Jiangyin People's Hospital, Wuxi, Jiangsu
  - xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xuzhou coal mining group General Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University（Department of Neurology ward 1）, Xuzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University（Department of Neurology ward 2）, Xuzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - The fourth peoples hospital of zhenjiang city, Zhenjiang, Jiangsu
  - Ganzhou city people's Hospital, Ganzhou, Jiangxi
  - The First People's Hospital of Jingdehzne City, Jingdezhen, Jiangxi
  - Affiliated Hospital of Jiujiang College, Jiujiang, Jiangxi
  - Jiujiang first people's Hospital, Jiujiang, Jiangxi
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Shangrao City People's Hospital, Shangrao, Jiangxi
  - Sino-Japanese Friendship Hospital Of Jilin University, Changchun, Jilin
  - The First Hospital Of Jilin University, Changchun, Jilin
  - Jilin Provincial People's Hospital, Changchun, Jilin
  - Xinhua Hospital affiliated to Dalian University, Dalian, Liaoning
  - Second People's Hospital of Huludao City, Huludao, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - First People's Hospital of Shenyang, Shenyang, Liaoning
  - Guyuan people's hospital, Guyuan, Ningxia
  - The Fifth People's Hospital of Ningxia Hui Autonomous Region, Shizuishan, Ningxia
  - The Second People's Hospital of Shizuishan, Shizuishan, Ningxia
  - Shizuishan First People's Hospital, Shizuishan, Ningxia
  - Second people's Hospital of shizuishan, Shizuishan, Ningxia
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Yinchuan First People's Hospital, Yinchuan, Ningxia
  - Cardiovascular and Cerebrovoscular Hospital of General Hospital of Ningxia Med. Univ, Yinchuan, Ningxia
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Zhongwei People's Hospital, Zhongwei, Ningxia
  - Baoji High-tech People's Hospital, Baoji, Shaanxi
  - weinan Central Hospital, Weinan, Shaanxi
  - Xi 'an Hi-tech Hospital, Xi'an, Shaanxi
  - Xi 'an Fengcheng Hospital, Xi'an, Shaanxi
  - Xian 141 Hospital, Xi'an, Shaanxi
  - Dezhou People's Hospital, Dezhou, Shandong
  - Ningjin County People's Hospital, Dezhou, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Liaocheng City Third People's Hospital, Liaocheng, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Liaocheng Veterans Hospital, Liaocheng, Shandong
  - The Brain Hospital of Liaocheng People's Hospital, Liaocheng, Shandong
  - Guanxian People's Hospital, Liaocheng, Shandong
  - Liaocheng City Second People's Hospital, Liaocheng, Shandong
  - Dongchangfu people's Hospital, Liaocheng, Shandong
  - Liaocheng Central Hospital, Liaocheng, Shandong
  - Linqing People's Hospital, Linqing, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Affiliated Hospital of Qingdao University Medical College, Qingdao, Shandong
  - Qingdao West Coast New Area People's Hospital, Qingdao, Shandong
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Sunshine Union Hospital, Weifang, Shandong
  - weihai Central Hospital, Weihai, Shandong
  - Wendeng District People's Hospital, Weihai, Shandong
  - Penglai People's Hospital, Yantai, Shandong
  - Yantai Beihai Hospita, Yantai, Shandong
  - Putuo District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai 7th People's Hospital, Shanghai, Shanghai Municipality
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Heping Hospital affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Datong Fifth People's Hospital, Datong, Shanxi
  - The Third People's Hospital of Datong, Datong, Shanxi
  - Shanxi cardiovascular disease hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Taiyuan Iron and Steel (Group) Co, Ltd,General Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Xi 'an First Hospital, Xi’an, Shanxi
  - Shenzhen Integrated Chinese and Western Medicine Hospital, Shenzhen, Shenzhen
  - Shenzhen Luohu People's Hospital, Shenzhen, Shenzhen
  - Shenzhen Second People's Hospital, Shenzhen, Shenzhen
  - Huazhong University of Science and Technology Union Shenzhen Hospital, Shenzhen, Shenzhen
  - West China Hospital Of Sichuan University, Chengdou, Sichuan
  - Chengdu second Municipal People'sHospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - dazhou Central Hospital, Dazhou, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Guiyang, Xinjiang Autonomous Region
  - People's Hospital Of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang Autonomous Region
  - Friendship Hospital of Ili Kazak Autonomous Prefecture, Yining, Xinjiang Autonomous Region
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Hangzhou first people's Hospital, Hangzhou, Zhejiang
  - lishui municipal Central Hospital, Lishui, Zhejiang
  - Zhejiang Wenzhou Medical College Third Affiliated Hospital, Ruian, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao J, Tian X, Yang X, Xu Q, Xia X, Zhang Y, Xie X, Bath PM, Jing J, Wang Y, Meng X, Wang A. Effect of insulin resistance on ticagrelor-versus clopidogrel-based dual antiplatelet therapy for secondary prevention of stroke in carriers of CYP2C19 loss-of-function mutations. CMAJ. 2026 Jan 18;198(2):E36-E43. doi: 10.1503/cmaj.241581. PMID 41554550
- [Derived] Lin J, Zhou H, Wang Y, Jin A, Li S, Zhang L, Meng X, Xie X, Jing J, Jiang Y, Wang Y, Zhao X, Li H, Li Z, Wang Y; CHANCE-2 Investigators. Lp-PLA2 Activity and Genotype-Guided Dual Antiplatelet Therapy in Minor Stroke or Transient Ischemic Attack. Stroke. 2026 Jan 13. doi: 10.1161/STROKEAHA.125.052954. Online ahead of print. PMID 41527826
- [Derived] Li H, Xia X, Xu Q, Meng X, Wang Y, Wang A. Differential Effect of Ticagrelor Versus Clopidogrel by Causative Classification of Stroke Classification and Vascular Cellular Adhesion Molecule-1 Level on the Risk of Recurrent Stroke: A Post Hoc Analysis of the CHANCE-2 Trial. J Am Heart Assoc. 2026 Jan 6;15(1):e042259. doi: 10.1161/JAHA.125.042259. Epub 2025 Dec 18. PMID 41413755
- [Derived] Feng Z, Zhang F, Jin A, Li X, Li Y, Chu Q, Xue J, Cheng A, Lin J, Li H, Meng X, Wang Y, Xu J. Genotype-guided dual antiplatelet therapy in minor stroke or transient ischemic attack with metabolic syndrome: A post hoc analysis of CHANCE-2. Diabetes Obes Metab. 2026 Jan;28(1):625-633. doi: 10.1111/dom.70243. Epub 2025 Oct 27. PMID 41145384
- [Derived] Lin X, Guo C, Meng X, Zhao X, Li H, Wang Y, Yang J. PCISOS Risk Profiles Stratify Heterogeneous Outcomes in Minor Posterior Circulation Ischemic Stroke: A Post Hoc Analysis of the CHANCE-2 Trial. Stroke. 2025 Dec;56(12):3371-3381. doi: 10.1161/STROKEAHA.125.053054. Epub 2025 Sep 10. PMID 40927840
- [Derived] Xie X, Jing J, Wang A, Xu Q, Zhao X, Lin J, Chen P, Jiang Y, Wang Y, Li H, Meng X, Wang Y. Dual antiplatelet therapy with ticagrelor vs clopidogrel in patients with TIA or minor stroke with or without symptomatic carotid artery stenosis: a post hoc analysis of the CHANCE-2 trial. Stroke Vasc Neurol. 2025 Oct 27;10(5):551-559. doi: 10.1136/svn-2024-003293. PMID 39773886
- [Derived] Xie X, Jing J, Meng X, Johnston SC, Bath PM, Li Z, Zhao X, Wang Y, Xu Q, Wang A, Jiang Y, Li H, Wang Y; CHANCE-2 Investigators. Dual Antiplatelet Therapy After Embolic Stroke of Undetermined Source: A Subgroup Analysis of the CHANCE-2 Trial. Stroke. 2024 Jul;55(7):1739-1747. doi: 10.1161/STROKEAHA.124.046834. Epub 2024 Jun 11. PMID 38860396
- [Derived] Wang A, Tian X, Xie X, Li H, Bath PM, Jing J, Lin J, Wang Y, Zhao X, Li Z, Liu L, Wang Y, Meng X. Differential effect of ticagrelor versus clopidogrel by homocysteine levels on risk of recurrent stroke: a post hoc analysis of the CHANCE-2 trial. CMAJ. 2024 Feb 11;196(5):E149-E156. doi: 10.1503/cmaj.231262. PMID 38346785
- [Derived] Zhang X, Jing J, Wang A, Xie X, Johnston SC, Li H, Bath PM, Xu Q, Lin J, Wang Y, Zhao X, Li Z, Jiang Y, Liu L, Chen W, Gong X, Li J, Han X, Meng X, Wang Y. Efficacy and safety of dual antiplatelet therapy in the elderly for stroke prevention: a subgroup analysis of the CHANCE-2 trial. Stroke Vasc Neurol. 2024 Nov 5;9(5):541-550. doi: 10.1136/svn-2023-002450. PMID 38286485
- [Derived] Meng X, Wang A, Tian X, Johnston C, Li H, Bath PM, Xu Q, Zhang Y, Xie X, Jing J, Lin J, Wang Y, Zhao X, Li Z, Jiang Y, Liu L, Wang Y. One-Year Outcomes of Early Therapy With Ticagrelor vs Clopidogrel in CYP2C19 Loss-of-Function Carriers With Stroke or TIA Trial. Neurology. 2024 Feb 13;102(3):e207809. doi: 10.1212/WNL.0000000000207809. Epub 2024 Jan 5. PMID 38181311
- [Derived] Wang A, Tian X, Xie X, Li H, Jing J, Lin J, Wang Y, Zhao X, Li Z, Liu L, Wang Y, Meng X. Effects of remnant cholesterol on the efficacy of genotype-guided dual antiplatelet in CYP2C19 loss-of -function carriers with minor stroke or transient ischaemic attack: a post-hoc analysis of the CHANCE-2 trial. EClinicalMedicine. 2023 Dec 2;67:102357. doi: 10.1016/j.eclinm.2023.102357. eCollection 2024 Jan. PMID 38125963
- [Derived] Wang C, Jia W, Jing J, Meng X, Wang A, Xu Q, Zhang X, Pan Y, Xie X, Johnston SC, Bath PM, Lin J, Jiang Y, Li H, Wang Y, Zhao X, Liu L, Li Z, Wang Y; CHANCE-2 Investigators. Ticagrelor Versus Clopidogrel in Minor Stroke or Transient Ischemic Attack With Intracranial Artery Stenosis: A Post Hoc Analysis of CHANCE-2. J Am Heart Assoc. 2023 Nov 7;12(21):e031611. doi: 10.1161/JAHA.123.031611. Epub 2023 Oct 27. PMID 37889172
- [Derived] Xie X, Jing J, Meng X, Claiborne Johnston S, Bath PM, Li Z, Zhao X, Liu L, Wang Y, Xu Q, Wang A, Jiang Y, Li H, Wang Y; CHANCE-2 Investigators. Dual Antiplatelet Therapies and Causes in Minor Stroke or Transient Ischemic Attack: A Prespecified Analysis in the CHANCE-2 Trial. Stroke. 2023 Sep;54(9):2241-2250. doi: 10.1161/STROKEAHA.122.042233. Epub 2023 Aug 7. PMID 37548009
- [Derived] Zhang J, Wang A, Tian X, Meng X, Xie X, Jing J, Lin J, Wang Y, Li Z, Liu L, Li H, Jiang Y, Zhao X, Wang Y. Impact of body mass index on efficacy and safety of ticagrelor versus clopidogrel in patients with minor stroke or transient ischemic attack. CMAJ. 2023 Jul 10;195(26):E897-E904. doi: 10.1503/cmaj.230262. PMID 37429630
- [Derived] Xie X, Johnston SC, Wang A, Xu Q, Bath PM, Pan Y, Li H, Lin J, Wang Y, Zhao X, Li Z, Jiang Y, Liu L, Xu A, Jing J, Meng X, Wang Y. Association of CYP2C19 Loss-of-Function Metabolizer Status With Stroke Risk Among Chinese Patients Treated With Ticagrelor-Aspirin vs Clopidogrel-Aspirin: A Prespecified Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2317037. doi: 10.1001/jamanetworkopen.2023.17037. PMID 37279000
- [Derived] Liu H, Jing J, Wang A, Xu Q, Meng X, Li H, Li Z, Wang Y. Stroke Recurrence and Antiplatelets in Posterior Versus Anterior Circulation Minor Stroke or Transient Ischemic Attack. Stroke. 2023 Apr;54(4):964-972. doi: 10.1161/STROKEAHA.122.041738. Epub 2023 Feb 15. PMID 36789773
- [Derived] Jing J, Xie X, Johnston SC, Bath PM, Li Z, Zhao X, Liu L, Wang Y, Xu Q, Wang A, Jiang Y, Li H, Meng X, Wang Y; CHANCE-2 Investigators. Genotype-Guided Dual Antiplatelet Use for Transient Ischemic Attack and Minor Stroke by Imaging Status: Subgroup Analysis of the CHANCE-2 Trial. Ann Neurol. 2023 Apr;93(4):783-792. doi: 10.1002/ana.26589. Epub 2023 Jan 20. PMID 36571569
- [Derived] Wang A, Meng X, Tian X, Zuo Y, Bath PM, Li H, Xie X, Jing J, Lin J, Wang Y, Zhao X, Liu L, Li Z, Jiang Y, Xu J, Wang F, Chen W, Cao M, Li J, Wang Y. Ticagrelor Aspirin vs Clopidogrel Aspirin in CYP2C19 Loss-of-Function Carriers With Minor Stroke or TIA Stratified by Risk Profile. Neurology. 2023 Jan 31;100(5):e497-e504. doi: 10.1212/WNL.0000000000201454. Epub 2022 Dec 19. PMID 36535779
- [Derived] Wang A, Xie X, Tian X, Johnston SC, Li H, Bath PM, Zuo Y, Jing J, Lin J, Wang Y, Zhao X, Li Z, Jiang Y, Liu L, Meng X, Wang Y. Ticagrelor-Aspirin Versus Clopidogrel-Aspirin Among CYP2C19 Loss-of-Function Carriers With Minor Stroke or Transient Ischemic Attack in Relation to Renal Function: A Post Hoc Analysis of the CHANCE-2 Trial. Ann Intern Med. 2022 Nov;175(11):1534-1542. doi: 10.7326/M22-1667. Epub 2022 Nov 1. PMID 36315949
- [Derived] Wang A, Meng X, Tian X, Johnston SC, Li H, Bath PM, Zuo Y, Xie X, Jing J, Lin J, Wang Y, Zhao X, Li Z, Jiang Y, Liu L, Wang F, Wang Y, Huang P, Chen G, Wang Y; CHANCE-2 Investigators. Effect of Hypertension on Efficacy and Safety of Ticagrelor-Aspirin Versus Clopidogrel-Aspirin in Minor Stroke or Transient Ischemic Attack. Stroke. 2022 Sep;53(9):2799-2808. doi: 10.1161/STROKEAHA.122.038662. Epub 2022 Jun 3. PMID 35656824
- [Derived] Wang Y, Meng X, Wang A, Xie X, Pan Y, Johnston SC, Li H, Bath PM, Dong Q, Xu A, Jing J, Lin J, Niu S, Wang Y, Zhao X, Li Z, Jiang Y, Li W, Liu L, Xu J, Chang L, Wang L, Zhuang X, Zhao J, Feng Y, Man H, Li G, Wang B; CHANCE-2 Investigators. Ticagrelor versus Clopidogrel in CYP2C19 Loss-of-Function Carriers with Stroke or TIA. N Engl J Med. 2021 Dec 30;385(27):2520-2530. doi: 10.1056/NEJMoa2111749. Epub 2021 Oct 28. PMID 34708996
- [Derived] Wang Y, Johnston C, Bath PM, Meng X, Jing J, Xie X, Wang A, Pan Y, Xu A, Dong Q, Wang Y, Zhao X, Li Z, Li H; CHANCE-2 Investigators. Clopidogrel with aspirin in High-risk patients with Acute Non-disabling Cerebrovascular Events II (CHANCE-2): rationale and design of a multicentre randomised trial. Stroke Vasc Neurol. 2021 Jun;6(2):280-285. doi: 10.1136/svn-2020-000791. Epub 2021 May 5. PMID 33952670